CLINICAL TRIAL: NCT05590715
Title: International, Multicentric, Observational Study to Characterize Subpopulations of Patients With Autism Spectrum Disorder
Brief Title: International Multicentric Observational Study to Characterize Subpopulations of Patients With Autism Spectrum Disorder
Status: Recruiting | Type: Observational
Sponsor: Stalicla SA (Industry)
Responsible Party: Sponsor
Other Study IDs: STA-B-001
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — DNA and RNA extraction, plasma and PBMC isolation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine sufficient number of biological and clinical markers to identify subgroups of potential best responders to a specific medication

ELIGIBILITY:
Inclusion Criteria:

* Participants previously diagnosed with ASD (DSM-5)
* Available well-documented health records within the first 2 years of life
* Participants must have a parent or reliable caregiver who agrees to provide information about the participant
* Participants willing and consenting or assenting to participate.

Exclusion Criteria:

* Episode of fever (i.e. ≥100.5 °F or ≥ 38 °C) or clinically significant illness without fever (as judged by the investigator), within 10 days before any study assessment.
* If the investigator assesses any unwillingness or any medical condition that may prevent the subject from completing this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female individuals with an autism diagnosis as defined by the DSM-5, adults (from 18 to 65 years of age, inclusive) and adolescents (from 12 to 17 years of age, inclusive).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characterisation of the ASD-Phen1 and ASD-Phen2 subpopulations. | Day 0
  A semi-structured medical questionnaire will be administered to collect clinical (sign and symptoms) and anthropomorphic features.
Molecular characterization of the ASD-Phen1 and ASD-Phen2 subpopulations | Day 0
  Better characterize subpopulations of ASD subjects and potentially identify/confirm a molecular signature specific of each subpopulation.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Fontoura, MD, PhD, Study Director — Stalicla SA
Locations (21):
- United States (9):
  - SARRC, Phoenix, Arizona
  - California Neuroscience Research, Sherman Oaks, California
  - BioPhase Research, Miami, Florida
  - The Angel Medical Research, Miami Lakes, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Missouri, Thompson Center for Autism & Neurodevelopmental Disorders, Columbia, Missouri
  - Golden Hearts Diagnostic, Alamogordo, New Mexico
  - Red Oak Psychiatry Associates, Houston, Texas
  - Alpine Research Organization, Clinton, Utah
- Australia (5):
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Locuspsych, Melbourne, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
- Spain (7):
  - Hospital General Universitario Dr Balmis, Alicante
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Infantil Universitario Nino Jesus (HIUNJS), Madrid
  - Hospital universitario Infanta Leonor, Madrid
  - Hospital Universitario Puerta De Hierro Majadahonda, Majadahonda
  - Policlina Gipuzkoa, San Sebastián
  - Hospital Álvaro Cunqueiro, Vigo